CLINICAL TRIAL: NCT00614523
Title: A Randomized, Double Blind, Placebo Controlled Study Evaluating the Efficacy and Safety of Romiplostim Treatment of Thrombocytopenia in Subjects With Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Brief Title: Romiplostim Treatment of Thrombocytopenia in Subjects With Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20060198
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: MDS; Myelodysplastic Syndromes; Thrombocytopenia
Keywords: MDS; Low Risk MDS; Intermediate-1 Risk MDS; Thrombocytopenia
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Romiplostim (Experimental): Weekly subcutaneous dosing based on platelet count for 26 weeks during the Test Treatment Period and for 24 weeks during the Extended Treatment Period, separated by a 4-week interim washout period. Starting dose is at 750 μg, up to a maximum dose of 1000 μg, or reduced to a minimum of 250 μg.
  Interventions: Biological: Romiplostim
- Placebo (Placebo Comparator): Weekly subcutaneous dosing with blinded matching placebo dose level for 26 weeks during the Test Treatment Period and for 24 weeks during the Extended Treatment Period, separated by a 4-week interim washout period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo is supplied in a 5 mL single use glass vial as a sterile, white, preservative-free, lyophilized powder.
  Arms: Placebo
Biological: Romiplostim — Romiplostim is supplied in a 5 mL single use glass vial as a sterile, white, preservative-free, lyophilized powder.
  Arms: Romiplostim

SUMMARY:
The Data Monitoring Committee (DMC) for study 20060198 recommended that all subjects discontinue treatment of study drug and continue to be followed for long term follow-up. Amgen adopted the DMC recommendation.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double blind, placebo controlled study designed to assess the efficacy and safety of romiplostim (formerly, AMG 531) treatment in thrombocytopenic MDS patients. The study is composed of a 26-week placebo controlled test treatment period (romiplostim versus Placebo), a 4 week interim wash-out period, a 24-week placebo controlled extended treatment period, and a 4-week follow-up period followed by an End of Study (EOS) visit. During the interim wash-out period, a bone marrow biopsy will be performed in the absence of growth factor to assess changes in the marrow. In the extended treatment period, safety assessments will continue and participants will be allowed to receive any standard of care treatments for MDS. Patients will be followed for survival for an additional 60 months following the End of Study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria: • Diagnosis of MDS using the World Health Organization (WHO) classification for myeloid neoplasms as assessed during the screening period. • Per MDS International Prognostic Scoring System (IPSS), low or intermediate-1 risk MDS as assessed during the screening period. • Mean of the 2 platelet counts taken within 4 weeks prior to randomization must be: - ≤ 20 x 10^9/L, (with no individual count >30 x 10^9/L during the screening period), with or without history of bleeding associated with diagnosis of MDS, OR - ≤ 50 x 10^9/L, (with no individual count >60 x 10^9/L during the screening period) with a history of bleeding associated with the diagnosis of MDS. • Patients must be ≥18 and ≤ 90 years of age at time of informed consent. Patients between 85 and 90 years of age must have been diagnosed with MDS ≤ 5 years from study start. • Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. • Adequate liver function, as evidenced by alanine aminotransferase (ALT) ≤ 3 times laboratory normal range, aspartate aminotransferase (AST) ≤ 3 times laboratory normal range and total bilirubin ≤ 2.0 times laboratory normal range. (Adequate liver function for patients with confirmed diagnosis of Gilbert's Disease evidenced by ALT ≤ 3 times laboratory normal range, and AST ≤ 3 times laboratory normal range.) • Serum creatinine concentration ≤ 2 mg/dl (≤176.8 μmol/L). • Bone marrow biopsy and aspirate with cytogenetics within 3 months of starting first dose of investigational product. • Written Informed Consent. Exclusion Criteria: • Have ever received any disease-modifying treatment for MDS. • Previously diagnosed with intermediate-2 or high risk MDS using the IPSS. • Prior history of leukemia, aplastic anemia, or other non-MDS related bone marrow stem cell disorder. • Prior history of hematopoietic stem cell transplantation. • Persistent peripheral blood monocytosis (≥ 3 months with an absolute monocyte count >1,000/μL) or known diagnosis of Chronic Myelomonocytic Leukemia per French-American-British Classification System for MDS (FAB) criteria. • Prior malignancy (other than in situ cervical cancer, non-melanoma skin cancer, or in situ carcinoma) unless treated with curative intent and without evidence of disease for ≥ 3 years before randomization. • Active or uncontrolled infections. • Unstable angina, congestive heart failure (New York Heart Association [NYHA] > class II), uncontrolled hypertension (diastolic >100 mmHg), uncontrolled cardiac arrhythmia, or recent (within 1 year) myocardial infarction. • History of arterial thrombosis (eg, stroke or transient ischemic attack) within the past year. • History of venous thrombosis that currently requires anti-coagulation therapy. • Received Interleukin (IL)-11 within 4 weeks of first dose of investigational product. • Have previously received any thrombopoietic growth factor. • Receipt of granulocyte-colony stimulating factor, (G-CSF), pegylated-G-CSF, or granulocyte macrophage-colony stimulating factor (GM-CSF) within 4 weeks of first dose of investigational product. • Planned receipt of peg-G-CSF or GM-CSF after first dose of investigational product. • Pregnant or breast feeding. • Patients of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator. Amgen recommends double barrier contraception is used for all applicable patients enrolled on this study. A double barrier method is defined as two methods of contraception, for example 2 actual barrier methods, or one actual barrier method and one hormonal method. • Patient has known sensitivity to any recombinant E coli-derived product (eg, Infergen®, Neupogen®, Somatropin, and Actimmune). • Previously enrolled into the 20060198 study or another romiplostim study. • Inability to comply with study procedures. • Patient currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-07-21 (Actual); Primary Completion 2011-03-31 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Diao G, Zeng D, Hu K, Ibrahim JG. Modeling event count data in the presence of informative dropout with application to bleeding and transfusion events in myelodysplastic syndrome. Stat Med. 2017 Sep 30;36(22):3475-3494. doi: 10.1002/sim.7351. Epub 2017 May 30. PMID 28560768
- [Background] Kantarjian HM, Fenaux P, Sekeres MA, Szer J, Platzbecker U, Kuendgen A, Gaidano G, Wiktor-Jedrzejczak W, Carpenter N, Mehta B, Franklin J, Giagounidis A. Long-term follow-up for up to 5 years on the risk of leukaemic progression in thrombocytopenic patients with lower-risk myelodysplastic syndromes treated with romiplostim or placebo in a randomised double-blind trial. Lancet Haematol. 2018 Mar;5(3):e117-e126. doi: 10.1016/S2352-3026(18)30016-4. Epub 2018 Jan 26. PMID 29396092
- [Background] Giagounidis A, Mufti GJ, Fenaux P, Sekeres MA, Szer J, Platzbecker U, Kuendgen A, Gaidano G, Wiktor-Jedrzejczak W, Hu K, Woodard P, Yang AS, Kantarjian HM. Results of a randomized, double-blind study of romiplostim versus placebo in patients with low/intermediate-1-risk myelodysplastic syndrome and thrombocytopenia. Cancer. 2014 Jun 15;120(12):1838-46. doi: 10.1002/cncr.28663. Epub 2014 Apr 4. PMID 24706489
- [Background] Platzbecker U, Sekeres MA, Kantarjian H, Giagounidis A, Mufti GJ, Jia C, Yang AS, Fenaux P. Relationship of different platelet response criteria and patient outcomes in a romiplostim myelodysplastic syndromes trial. Leukemia. 2014 Dec;28(12):2418-21. doi: 10.1038/leu.2014.253. Epub 2014 Sep 2. No abstract available. PMID 25179731
- [Background] Sekeres MA, Giagounidis A, Kantarjian H, Mufti GJ, Fenaux P, Jia C, Yang AS, Platzbecker U. Development and validation of a model to predict platelet response to romiplostim in patients with lower-risk myelodysplastic syndromes. Br J Haematol. 2014 Nov;167(3):337-45. doi: 10.1111/bjh.13037. Epub 2014 Jul 14. PMID 25039607
- [Background] Diao G, Zeng D, Hu K, Ibrahim JG. Semiparametric frailty models for zero-inflated event count data in the presence of informative dropout. Biometrics. 2019 Dec;75(4):1168-1178. doi: 10.1111/biom.13085. Epub 2019 Sep 2. PMID 31106400
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 21 July 2008, Last Subject Enrolled: 16 December 2010.
Period: Overall Study
Arm/Group | Placebo | Romiplostim
Started | 83 | 167
Completed | 20 | 36
Not Completed | 63 | 131
Not completed — Adverse Event | 4 | 20
Not completed — Death | 5 | 8
Not completed — Lack of Efficacy | 9 | 11
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 12 | 22
Not completed — Other | 6 | 11
Not completed — Ineligibility Determined | 1 | 2
Not completed — Disease Progression | 0 | 8
Not completed — Administrative Decision | 23 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romiplostim | Total
Number analyzed (Participants) | 83 | 167 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11.5) | 68.4 (12) | 67.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 72 | 102
  Male | 53 | 95 | 148
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 79 | 156 | 235
  Black or African American | 0 | 1 | 1
  Hispanic or Latino | 1 | 4 | 5
  Asian | 1 | 1 | 2
  Other | 2 | 5 | 7
Myelodysplastic Syndromes World Health Organization Classification [Number; unit: Participants] — RA: Refractory Anemia RAEB-1: Refractory Anemia with Excess Blasts-1 RAEB-2: Refractory Anemia with Excess Blasts-2 RARS: Refractory Anemia with Ringed Sideroblasts RCMD: Refractory cytopenia with multilineage dysplasia RCMD-RS: Refractory cytopenia with multilineage dysplasia and ringed sideroblasts MDS-U: Myelodysplastic syndrome - unclassified MDS associated with isolated del(5q).
  Participants
    RA | 5 | 6 | 11
    RARS | 0 | 2 | 2
    RAEB-1 | 9 | 24 | 33
    RAEB-2 | 0 | 1 | 1
    RCMD | 55 | 114 | 169
    RCMD-RS | 2 | 4 | 6
    MDS-U | 12 | 16 | 28
    MDS associated with isolated del 5Q | 0 | 0 | 0
Prior MDS Therapy [Number; unit: Participants] — Had received MDS therapy prior to enter the study
  Participants
    No | 70 | 133 | 203
    Yes | 13 | 34 | 47
Baseline Platelet Counts [Mean (Standard Deviation); unit: 10^9/L] | 21.5 (13) | 22.3 (11.5) | 22.0 (12.0)
International Prognostic Scoring System (IPSS) Total Score [Number; unit: Participants] — The IPSS uses three "prognostic indicators" to develop a "score" which may be useful in understanding how the MDS may progress:
  * the proportion of blast cells in the marrow;
  * the type of chromosomal changes, if any, in the marrow cells;
  * the presence of one or more low blood cell counts (cytopenias). Scores are sorted into one of four risk categories: 0 = low risk; 0.5-1.0 = intermediate-1; 1.5-2.0 = intermediate-2; >2.5 = high risk.
  Participants
    0 | 23 | 40 | 63
    0.5 | 38 | 86 | 124
    1 | 20 | 34 | 54
    1.5 | 0 | 1 | 1
    Missing | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Significant Bleeding Events
Description: A clinically significant bleeding event is defined as any bleeding event of grade ≥ 2 per the modified World Health Organization (WHO) bleeding scale: • Grade 0 = no bleeding • Grade 1 = petechia or mucosal or retinal bleeding not requiring intervention • Grade 2 = melena, hematemesis, hematuria, hemoptysis • Grade 3 = bleeding required red cell transfusion • Grade 4 = retinal bleeding with visual impairment • Grade 5 = non-fatal cerebral bleeding • Grade 6 = fatal cerebral bleeding • Grade 7 = fatal non-cerebral bleeding. Bleeding events that continue for more than 7 days were counted as separate events every eighth day. Multiple events that arose from one organ system on one day were collapsed into one single event. Bleeding events with a start date between the first dose date and the last dose date of the test treatment period+7 days are included.
Time Frame: Test Treatment Period (Weeks 1-26)
Population: Full analysis set includes all randomized patients.
Measure: Number; unit: events
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
events | 116 | 178
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p = 0.13, Anderson-Gill model; Anderson-Gill model using the model-based variance estimate and stratified by the randomization stratification factors; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.66 to 1.05] — Romiplostim /Placebo

2. Secondary Outcome: Annualized Rate of Platelet Transfusion Events
Description: A discrete platelet transfusion is any number of platelet transfusion administered within a 3-day period. Transfusions administered more than 3 days apart are counted as separate events. Transfusion given in the absence of any bleeding, when platelet count is >10x10^9/L, is not counted as a platelet transfusion event. Events with start date between the first dose date and the last dose date of the test treatment period +7 days are included. Exposure adjusted event rate per 100 patient-years = (events / patient-years * 100). Patient Year = total patient years of exposure to investigational product during 26 weeks test treatment period.
Time Frame: Test Treatment Period (Weeks 1-26)
Population: Full analysis set includes all randomized patients.
Measure: Mean (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
events per 100 patient-years | 1013.5 [905.2 to 1131.3] | 748.9 [681.3 to 821.4]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p < 0.001, Poisson regression model; Poisson regression model with treatment and stratification factors as covariates; Risk Ratio (RR) = 0.766, 95% CI 2-sided [0.66 to 0.88] — Romiplostim /Placebo

3. Secondary Outcome: Annualized Rate of Overall Bleeding Events
Description: The time from first dose of study drug to the last dose of 26-week test treatment period. A bleeding event is defined as any bleeding event reported during the test treatment period. Bleeding events that continue for more than 7 days are counted as separate events every eighth day. Multiple events that arose from one organ system on one day are collapsed into one single event. Exposure adjusted event rate per 100 patient-years = events / patient-year * 100).
Time Frame: Test Treatment Period (Weeks 1-26)
Population: Full analysis set includes all randomized patients.
Measure: Mean (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
events per 100 patient-years | 3786.4 [3574.1 to 4008.0] | 3459.9 [3312.8 to 3611.9]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p = 0.026, Poisson regression model; Poisson regression model with treatment and stratification factors as covariates; Risk Ratio (RR) = 0.922, 95% CI 2-sided [0.86 to 0.99] — Romiplostim /Placebo

4. Secondary Outcome: Annualized Rate of Total Platelet Transfusion Units
Description: The time from first dose of study drug to the last dose of 26-week test treatment period. A unit of platelets is defined as a single pack of pooled platelet-rich plasma comprised of 6 to 8 individual platelet concentrate packs (200 to 400 mL), a single pack of pooled buffy-coat concentrate, or 1 apheresis (single donor) concentrate. Exposure adjusted event rate per 100 patient-years = events / patient-years * 100.
Time Frame: Test Treatment Period (Weeks 1-26)
Population: Full analysis set includes all randomized subjects
Measure: Mean (95% Confidence Interval); unit: units per 100 patient-years
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
units per 100 patient-years | 3120.2 [2927.8 to 3322.0] | 2221.8 [2104.2 to 2344.2]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p < 0.001, Poisson Regression model; Poisson regression model with treatment and stratification factors as covariates; Risk Ratio (RR) = 0.739, 95% CI 2-sided [0.68 to 0.8] — Romiplostim /Placebo

5. Secondary Outcome: Number of Participants With Platelet Hematologic Improvement (HI-P)
Description: Platelet Hematologic Improvemen defined by the international working group (IWG) as: an absolute increase in platelet count of ≥ 30 x 10^9/L for a patient starting with a platelet count of ≥ 20 x 10^9/L or an increase in platelet count from < 20 x 10^9/L to ≥ 20 x 10^9/L and by at least 100% in a patient that started with a platelet count < 20 x 10^9/L. To account for any possible contribution from platelet transfusions, platelet counts within 3 days following administration of platelet transfusion is not counted towards the platelet hematologic improvement endpoint. If no platelet measurements are available on the weekly scheduled dose day, then that week is not counted towards the platelet hematologic improvement endpoint.
Time Frame: Test Treatment Period (Weeks 1-26)
Population: Full analysis set includes all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
Participants | 3 | 61
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test controlling for stratification factors; Odds Ratio (OR) = 15.6, 95% CI 2-sided [4.7 to 51.8] — Romiplostim /Placebo

6. Secondary Outcome: Exposure-adjusted Total Duration of Platelet Hematologic Improvement (HI-P) in the Absence of Platelet Transfusions
Description: Duration for participants who did not report HI-P during the period is 0. A platelet hematologic improvement (HI-P) is defined by an MDS International Working criteria as patients with a baseline platelet count of ≥ 20 x 10^9/L achieving an absolute increase of ≥ 30 x 10^9/L or increasing the platelet count to above 20 x 10^9/L and by at least 100% in patients with a baseline of < 20 x 10^9/L for at least 8 consecutive weeks. To account for any possible contribution from platelet transfusions, platelet counts within 3 days following administration of platelet transfusion is not counted towards the platelet hematologic improvement endpoint. If no platelet measurements are available on the weekly scheduled dose day, then that week is not counted towards the platelet hematologic improvement endpoint. The durations of HI-P are cumulative if more than one incidence occurred. Exposure adjusted event rate per 100 patient-weeks = total number of weeks / patient-weeks * 100.
Time Frame: Test Treatment Period (Weeks 1-26)
Population: Full analysis set includes all randomized patients.
Measure: Mean (95% Confidence Interval); unit: weeks per 100 patient-weeks
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
weeks per 100 patient-weeks | 2.57 [1.85 to 3.47] | 35.02 [32.98 to 37.16]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p = 0.032, Poisson regression model; Poisson regression model with treatment and stratification factors as covariates; Risk Ratio (RR) = 1.402, 95% CI 2-sided [1.03 to 1.91] — Romiplostim /Placebo

7. Secondary Outcome: Number of Participants Who Died
Time Frame: From randomization to 58 weeks, the end of study visit or the closest available follow-up information up to 58 weeks from the long term follow-up for those who discontinued the study early, with a data cut-off date of 20 July 2012.
Population: Full analysis set includes all randomized patients.
Measure: Number; unit: participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
participants | 17 [NA to NA] | 30 [NA to NA]

8. Secondary Outcome: Time to Death
Description: Overall survival was calculated using Kaplan-Meier methods. For patients who discontinued early, additional information from the long term follow-up are added (closest available follow-up information up to 58 weeks).
Time Frame: as for outcome 7
Population: Full analysis set includes all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
months | NA [NA to NA] — Median and confidence intervals were not estimable due to the low number of deaths. | NA [NA to NA] — Median and confidence intervals were not estimable due to the low number of deaths.

9. Secondary Outcome: Kaplan-Meier Estimate of Survival at Month 12
Description: Overall survival was calculated using Kaplan-Meier methods.
Time Frame: Month 12, with a data cut-off date of 20 July 2012.
Population: Full analysis set includes all randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 83 | 167
percentage of participants | 78 [67 to 86] | 83 [76 to 88]

10. Secondary Outcome: Annualized Rate of Patient-reported Bleeding Events
Description: The number of bleeding events was obtained from the thrombocytopenia symptoms (Th-symptoms) survey. Patients reported spontaneous bleeding to have occurred 0, 1 or 2, 3 or 4, 5 or 6, or 7 or more times in the past week. The lower threshold of bleeding counts is used for conservative purposes (i.e., the "3" is used for the response option of "3 or 4 times"). Exposure adjusted event rate per 100 patient-years = number of events / patient-year * 100.
Time Frame: Test Treatment Period (Weeks 1-26)
Population: The Patient Reported Outcomes (PRO) analysis set consists of patients in the full analysis set who also completed the baseline and at least one post-baseline assessment for any PRO measure.
Measure: Mean (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 82 | 162
events per 100 patient-years | 1995 [1840.5 to 2158.9] | 1264 [1175.1 to 1357.7]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p < 0.001, Poisson regression model; Poisson regression model with treatment and stratification factors as covariates; Risk Ratio (RR) = 0.639, 95% CI 2-sided [0.57 to 0.71] — Romiplostim /Placebo

ADVERSE EVENTS:
Time Frame: 58 weeks
Description: The safety analysis set consisted of 250 patients including 168 in the romiplostim group and 82 in the placebo group. One patient enrolled in the placebo group received 1 dose of romiplostim at week 4 of the extended treatment period. Results for this patient were analyzed as part of the romiplostim group in the Safety Analysis Set.
Arm/Group | Placebo | Romiplostim
Serious Adverse Events (participants affected / at risk) | 22/82 | 67/168
Other Adverse Events (participants affected / at risk) | 74/82 | 146/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Romiplostim (N=168)
Anaemia (Blood and lymphatic system disorders) | 2 | 7
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 5
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2
Retinal detachment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 7
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 1 | 2
Chronic sinusitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia sepsis (Infections and infestations) | 1 | 0
External ear cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gingival infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 8
Pneumonia viral (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Urosepsis (Infections and infestations) | 0 | 1
Viral pericarditis (Infections and infestations) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 4
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Blast cell count increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Myeloblast count increased (Investigations) | 0 | 2
Oxygen saturation decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2
Encephalitis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Wallenberg syndrome (Nervous system disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Romiplostim (N=168)
Anaemia (Blood and lymphatic system disorders) | 7 | 16
Conjunctival haemorrhage (Eye disorders) | 5 | 9
Abdominal pain (Gastrointestinal disorders) | 5 | 10
Constipation (Gastrointestinal disorders) | 6 | 9
Diarrhoea (Gastrointestinal disorders) | 10 | 23
Gingival bleeding (Gastrointestinal disorders) | 14 | 33
Mouth haemorrhage (Gastrointestinal disorders) | 8 | 21
Nausea (Gastrointestinal disorders) | 7 | 27
Vomiting (Gastrointestinal disorders) | 5 | 8
Asthenia (General disorders) | 6 | 22
Fatigue (General disorders) | 7 | 24
Injection site haematoma (General disorders) | 11 | 12
Oedema peripheral (General disorders) | 7 | 26
Pyrexia (General disorders) | 12 | 17
Vessel puncture site haematoma (General disorders) | 6 | 6
Nasopharyngitis (Infections and infestations) | 8 | 14
Oral herpes (Infections and infestations) | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 6 | 6
Contusion (Injury, poisoning and procedural complications) | 10 | 41
Decreased appetite (Metabolism and nutrition disorders) | 2 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 17
Dizziness (Nervous system disorders) | 6 | 16
Headache (Nervous system disorders) | 10 | 29
Syncope (Nervous system disorders) | 5 | 0
Insomnia (Psychiatric disorders) | 2 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32 | 66
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Blood blister (Skin and subcutaneous tissue disorders) | 11 | 25
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 | 20
Petechiae (Skin and subcutaneous tissue disorders) | 20 | 42
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 10
Rash (Skin and subcutaneous tissue disorders) | 10 | 12
Capillary fragility (Vascular disorders) | 5 | 0
Haematoma (Vascular disorders) | 33 | 58
Haemorrhage (Vascular disorders) | 15 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial resul